CLINICAL TRIAL: NCT03282487
Title: Optimising Steroid Replacement in Patients With Adrenal Insufficiency
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The Adelaide and Meath Hospital, incorporating The National Children's Hospital (Other)
Responsible Party: Principal Investigator, Dr Mark Sherlock, Consultant Endocrinologist, The Adelaide and Meath Hospital, incorporating The National Children's Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2016/09/05
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Adrenal Insufficiency
Keywords: cortisol; adrenal insufficiency; hypopituitarism; hydrocortisone
MeSH Terms: conditions — Adrenal Insufficiency; Hypopituitarism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional immediate release hydrocortisone (No Intervention)
- Modified release Hydrocortisone (Active Comparator): 12 weeks of modified release hydrocortisone (Plenadren)
  Interventions: Drug: Modified release hydrocortisone
- Healthy control group (No Intervention): Same research laboratory measurements performed in a healthy control group for comparison to patient group

INTERVENTIONS:
Drug: Modified release hydrocortisone — Patients will switch from their usual conventional immediate release hydrocortisone to daily dose equivalent of modified release hydrocortisone (Plenadren®)
  Other Names: Plenadren
  Arms: Modified release Hydrocortisone

SUMMARY:
Adrenal insufficiency is a condition where the adrenal glands do not produce an adequate amount of steroid hormones. The aetiology of adrenal insufficiency can be primary or secondary. Patients will adrenal insufficiency have increased morbidity and mortality. In recent years there has been concern regarding what is the optimal dose and regimen of steroid replacement for patients. Unfortunately there is no accurate way of monitoring if a patient is on too much or too little steroid. We have shown in hypopituitary patients with secondary adrenal insufficiency that higher doses of hydrocortisone may be harmful. This reason for this is not fully understood.

In recent years, a modified release hydrocortisone tablet (Plenadren) taken once per day (unlike conventional immediate release hydrocortisone which requires twice or thrice daily regimen) has come on the market. This tablet has shown to a have a steroid profile that more closely resembles normal physiology, avoiding the peak steroid levels that occur during thrice daily regimens, which may be of importance for improving outcome in adrenal insufficiency patients. It also shown improved cardiovascular risk factors, glucose metabolism and quality of life in compared to conventional treatment.

The aim of our study is to assess the effect of hydrocortisone therapy on how the body uses and breaks down (metabolises) steroids. This will be done by several different research methods: by measuring markers of steroid action and metabolism in blood, urine and within the fat tissue under the skin in the abdomen. These results will be compared in the same patient while on their usual hydrocortisone and after switching to modified release hydrocortisone for 12 weeks, and to results from a normal healthy control group who are not on steroid replacement.

This will be the first study to assess the impact of this new modified release hydrocortisone in relation to tissue steroid metabolism. The results will potentially help us to improve the treatment of patients with steroid deficiency and reduce the side effects seen in these patients.

DETAILED DESCRIPTION:
This is a prospective, cross-over study. This study cannot be blinded or placebo controlled due to the risk of adrenal crisis in the study population with primary and secondary adrenal insufficiency.

The aim of study is to assess the effect of immediate release and modified release hydrocortisone therapy on corticosteroid metabolism and 11-HSD1 in vivo (by assessment of urine metabolites and liver/ adipose tissue metabolism) by using several translational research approaches. This will also be compared to normal healthy controls to assess which treatment protocol is most physiological.

Study Objectives

* To assess the effect of changing to modified release hydrocortisone therapy on global corticosteroid metabolism as assessed by urinary steroid metabolite profiles.
* To assess the effect of changing to modified release hydrocortisone therapy on adipose tissue corticosteroid metabolism and action
* To assess the effect of changing to modified release hydrocortisone on hepatic corticosteroid metabolism.
* To assess the effect of changing to modified release hydrocortisone therapy on patient quality of life (QoL) as assessed through validated QoL questionnaires.
* To compare results to normal healthy controls to assess which treatment protocol is most physiological.
* To assess potential biomarkers for adequacy of hydrocortisone replacement therapy.

Patients will switch from their usual conventional immediate release hydrocortisone to daily dose equivalent of modified release hydrocortisone (Plenadren®) for 12 weeks.Other hormone replacement therapy regimens will not be adjusted during the study period.

Research laboratory measurements will be performed at baseline and 12 weeks of modified release hydrocortisone. At the end of the intervention treatment period, the patients will be shifted to their usual hydrocortisone treatment and will be followed at the outpatient clinic according to the directives of the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18years of age with Primary Adrenal Insufficiency (Addison's disease) confirmed on biochemical testing.
* Male or female patients ≥ 18years of age with ACTH deficiency defined by a stimulated peak cortisol in response to insulin-induced hypoglycaemia or short synacthen testing <400 nmol/l, with known organic pituitary disease, and no adjustment in hormone replacement for at least 3 months prior to study entry.
* Signed informed consent to participate in the study

Exclusion Criteria:

* Age < 18 years
* Patients with acute medical or surgical illness
* Patients with advanced cardiac/pulmonary disease
* Patients with a terminal illness
* Patients on glucocorticoids for purposes other than ACTH deficiency
* Patients on agents that interfere with corticosteroid metabolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-09-05 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Global corticosteroid metabolism | At baseline and after 12 weeks of Plenadren(intervention) treatment
  Urinary steroid metabolite profiles.
Adipose tissue corticosteroid metabolism | At baseline and after 12 weeks of Plenadren(intervention) treatment
  Cortisol generation profile using adipose tissue microdialysis catheter
Hepatic corticosteroid metabolism | At baseline and after 12 weeks of Plenadren(intervention) treatment
  Serum Cortisol generation profile

SECONDARY OUTCOMES:
Quality of Life questionnaires | At baseline and after 12 weeks of Plenadren(intervention) treatment
Potential biomarkers for adequacy of hydrocortisone replacement | At baseline and after 12 weeks of Plenadren(intervention) treatment
  Gene and protein expression of adipose tissue samples

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sherlock, Principal Investigator — Adelaide and Meath Hospital incorporating the national childrens hospital, Tallaght, Dublin, Ireland
Locations (1):
- Adelaide and Meath Hospital incorporating the National Childrens Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dineen RA, Martin-Grace J, Ahmed KMS, Taylor AE, Shaheen F, Schiffer L, Gilligan LC, Lavery GG, Frizelle I, Gunness A, Garrahy A, Hannon AM, Methlie P, Eystein SH, Stewart PM, Tomlinson JW, Hawley JM, Keevil BG, O'Reilly MW, Smith D, McDermott J, Healy ML, Agha A, Pazderska A, Gibney J, Behan LA, Thompson CJ, Arlt W, Sherlock M. Tissue Glucocorticoid Metabolism in Adrenal Insufficiency: A Prospective Study of Dual-release Hydrocortisone Therapy. J Clin Endocrinol Metab. 2023 Nov 17;108(12):3178-3189. doi: 10.1210/clinem/dgad370. PMID 37339332